CLINICAL TRIAL: NCT00703456
Title: The Effect of Balance Training on Unloading Reaction in Individuals With Functional Ankle Instability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 10866
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Ankle Injury
Keywords: Functional ankle instability; Balance training
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Balance Training, 3 times a week for 4 weeks
  Interventions: Behavioral: Balance Training
- 2 (No Intervention): Education/No intervention

INTERVENTIONS:
Behavioral: Balance Training — balance training three days per week for 4 weeks during single limb standing
  Arms: 1

SUMMARY:
The aim of this study is to determine the effect of a balance training intervention on the change in hyper-reactivity to unloading reaction, ankle joint laxity, ankle joint proprioception and evertor muscle weakness in individuals with functional ankle instability (FAI) using quantitative biomechanical and neuromuscular measurements.

We hypothesize that experimental FAI group will demonstrate a significant decline in unloading reaction following balance training while FAI control group will not show a significant decline in unloading reaction without training. We further hypothesize that experimental FAI group will demonstrate a significant improvement in the FAI score after the balance training measured by Ankle Instability questionnaire. Following balance training, there will be a significant correlation between the change in FAI score and change in the unloading reaction in the experimental group.

DETAILED DESCRIPTION:
Conflicting results have been reported regarding the effect of ankle sprain on the proprioceptive sensation of the ankle, peroneal muscle strength and ankle joint laxity in the past research studies related to FAI. In spite of controversies regarding etiological factors for FAI, balance training has been widely used in sports medicine clinics to treat FAI. Most of these studies have focused on the identification of postural control deficits in patients with FAI rather than trying to understand the mechanism of balance training on etiological factors of FAI.

Hyper-reactivity of the ankle joint with FAI may be an important factor for the ankle "giving way" episode. Patients may develop injury-induced hyper-reactivity for unloading reaction through an adaptation to physical conditions of the ankle joint after injury. Clinical studies performed with selective nerve blocks along with electrophysiology studies performed in animals have led to the generally accepted conclusion that enhanced pain induced by peripheral nerve injury is associated with increased spontaneous and evoked discharges from injured and/or adjacent uninjured nerves. Persistent primary afferent inputs are believed to cause a state of central (i.e. "spinal") sensitization and enhancing responses to sensory inputs i.e. hyper-reactivity.

The ankle "giving way" is a complex phenomenon where any mechanical and neuromuscular factor or a combination of mechanical and neuromuscular factors may be at fault including ankle hyper-reactivity, joint laxity, proprioceptive deficit, and muscle weakness. The purpose of this study is to examine the effect of balance training intervention on the various etiological factors of FAI and to develop an objective measurement for physiological features related to FAI.

The study will help us to understand the mechanism of balance training on FAI and help us to determine the scope and limitations of balance training on FAI subjects in clinical settings to evaluate treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 45 years
* unilateral functional ankle instability (grade II or III)
* at least four weeks after acute lateral ankle sprain
* ongoing symptom of ankle "giving way" episode during functional activities
* active in exercise at least 2 hour per week
* seeking medical treatment for ankle symptoms
* being able to complete the test and training tasks.

Exclusion Criteria:

* severe ankle pain and swelling
* ankle surgery in either leg
* gross limitation in ankle range of motion
* lower extremity injury other than lateral ankle sprain in past 12 weeks, (5) current enrollment in formal rehabilitation program
* history of insulin-dependent diabetes
* any systemic disease that might interfere with sensory input or muscle function of the lower extremity
* any joint disease or bony fracture in the lower extremity
* any previous experience of intolerance to electrical stimulation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Vertical force variation | 6 weeks

SECONDARY OUTCOMES:
ankle inversion flexibility, ankle proprioception, ankle evertor strength, modified cumberland ankle instability tool questionnaire | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States